CLINICAL TRIAL: NCT01822288
Title: The Impact of Different Hormone Therapy Regimens on Lower Urinary Tract Symptoms, Sexual Function and Psychosomatic Disorder
Brief Title: The Impact of Hormone Therapy on Lower Urinary Tract Symptoms, Sexual Function and Psychosomatic Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Principal Investigator, Sheng-Mou Hsiao, Chief, Department of Obstetrics & Gynecology, Far Eastern Memorial Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 101080-F
Record Dates: First submitted 2012-11-26; First posted 2013-04-02 (Estimated); Last update posted 2022-02-23 (Actual); Status verified 2021-12

CONDITIONS: Menopausal Syndromes
Keywords: Menopause; Tibolone; Estradiol; Hormone therapy
MeSH Terms: interventions — tibolone; Lunelle

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tibolone group (Experimental): Tibolone (2.5 mg per day)for 12 consecutive weeks. Tibolone should be paid by patient herself, and does not cover by Taiwan Government health insurance.
  Interventions: Drug: Tibolone
- Conventional hormone therapy group (Active Comparator): Estradiol valerate (E2V) 1mg & medroxyprogesterone acetate (MPA) 2.5 mg per day for 12 consecutive weeks, and this drug is paid by Taiwan Government health care insurance.
  Interventions: Drug: Estradiol & medroxyprogesterone acetate

INTERVENTIONS:
Drug: Tibolone — Tibolone 2.5 mg once a day for patients with menopausal syndrome (self-paid)
  Arms: Tibolone group
Drug: Estradiol & medroxyprogesterone acetate — Estradiol & medroxyprogesterone acetate once a day for patients with menopausal syndromes, for patients without the need for self-paid drug
  Arms: Conventional hormone therapy group

SUMMARY:
Menopausal syndromes includes somatic symptom, psychosomatic symptoms, sexual dysfunction and even urinary symptoms. Hormone therapy (HT) is widely used for controlling menopausal symptoms. Common HT for menopausal syndrome with intact uterus includes tibolone, estradiol valerate (E2V) 1mg & medroxyprogesterone acetate (MPA) 2.5 mg, and conjugated equine estrogens & MPA.

However, only a few literatures mentioned about the therapeutic effect of tibolone, but lack of comparison research about their therapeutic effect on somatic symptoms, psychosomatic symptoms, sexual dysfunction and even urinary symptoms. The knowledge of the above therapeutic effects should be important for choosing a suitable medication. Therefore, the aim of this study is to assess the therapeutic effect on somatic symptoms, psychosomatic symptoms, sexual dysfunction and even urinary symptoms between tibolone and E2V/MPA.

ELIGIBILITY:
Inclusion Criteria:

* All female patients with intact uterus who seek for medical treatment for menopausal syndrome

Exclusion Criteria:

* patients with gynecologic or breast cancers

Ages: 40 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2012-11-16 (Actual); Primary Completion 2021-07-08 (Actual); Study Completion 2021-08-26 (Actual)

PRIMARY OUTCOMES:
Menopausal symptoms | 12 weeks
  To clarify any difference of reduction in menopausal symptom scores between these two groups

SECONDARY OUTCOMES:
sexual function | 12 weeks
  To clarify any difference of improvements of sexual function scores between these two groups
lower urinary tract symptoms | 12 weeks
  To clarify any difference of improvements of lower urinary tract symptoms scores between these two groups
psychosomatic symptoms | 12 weeks
  To clarify any difference of improvements of psychosomatic symptoms scores between these two groups

CONTACTS AND LOCATIONS:
Locations (1):
- Far Eastern Memorial Hospital, Banqiao District, New Taipei, Taiwan

REFERENCES:
- [Derived] Hsiao SM, Liao SC. Effect of tibolone vs hormone replacement therapy on climacteric symptoms and psychological distress. J Chin Med Assoc. 2024 Feb 1;87(2):189-195. doi: 10.1097/JCMA.0000000000001012. Epub 2023 Oct 26. PMID 37882059